CLINICAL TRIAL: NCT01569464
Title: A Phase 3B, Double-Blind, Randomized, Placebo-Controlled Study of Rotigotine and Its Effect on All-Day Functioning and Quality of Life in Subjects With Moderate to Severe Idiopathic Restless Legs Syndrome
Brief Title: Rotigotine Effect on All-day Functioning and Quality of Life in Subjects With Moderate to Severe Restless Legs Syndrome (RLS)
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RL0003
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Restless Legs Syndrome; Neupro®
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Active Comparator): Rotigotine patches titrated from 1 mg/ 24 hr - 3 mg /24 hr or until effective or maximum dose is reached.
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo patches titrated from 1 mg/ 24 hr - 3 mg/ 24 hr or until effective or maximum dose was reached.
  Placebo 1 mg/ 24 hr, Placebo 2 mg/ 24 hr, Placebo 3 mg/ 24 hr, one patch every 24 hours
  7 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rotigotine — Transdermal patch containing Rotigotine formulated in an adhesive matrix. Subjects were to be treated with their optimal dose which consisted of one of the dose strengths below:
  Rotigotine 1 mg /24 hr, Rotigotine 2 mg/ 24 hr, Rotigotine 3 mg/ 24 hr, One patch every 24 hours
  7 weeks (titration plus maintenance)
  Other Names: Neupro®
  Arms: Rotigotine
Other: Placebo — Placebo patches titrated from 1 mg/ 24 hr - 3 mg/ 24 hr or until effective or maximum dose was reached.
  Placebo 1 mg/ 24 hr, Placebo 2 mg/ 24 hr, Placebo 3 mg/ 24 hr, one patch every 24 hours.
  7 weeks (titration plus maintenance)
  Arms: Placebo

SUMMARY:
The purpose of the study is to show that Rotigotine improves Restless Legs Syndrome (RLS) symptoms in subjects with moderate to severe RLS during both day and evening.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)-approved written Informed Consent Form (ICF) is signed and dated by the subject
* Subject understands the investigational nature of the study and is willing and able to comply with the study requirements. Subject is willing to accept that he/she might be treated with Placebo during the Treatment Period
* Subject is male or female, and is ≥ 18 and ≤ 75 years of age
* Subject is able to apply/remove the study patch correctly
* Subject meets the diagnosis of Idiopathic Restless Legs Syndrome (IRLS) based on the 4 essential clinical features according to the International Restless Legs Syndrome Study Group (Allen et al, 2003):
* 1. An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs. (The urge to move can be present without uncomfortable sensations. Arms or other body parts can also be affected)
* 2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying down or sitting
* 3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues
* 4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night. (When symptoms are very severe, the worsening at night may not be noticeable but must have been previously present)
* At Baseline (Visit 2), subject has a score of ≥ 11 on the RLS-Diagnostic Index (RLS-DI) (Benes and Kohnen, 2009)
* Subject must attempt all 4 Suggested Immobilization Test (SIT) assessments at Baseline (Visit 2)
* At Baseline (Visit 2) subject has an average Multiple Suggested Immobilization Test Discomfort Scale (m-SIT-DS) of at least 1.5 over the course of the Multiple Suggested Immobilization Test (m SIT)
* The subject's Body Mass Index is ≥ 18 kg/m^2 and ≤ 35 kg/m^2 at Visit 1
* At Baseline (Visit 2), subject has a score of ≥ 15 on the International Restless Legs Scale (IRLS) (indicating moderate to severe RLS)
* At Baseline (Visit 2), subject has a score of "Severe" or "Very Severe" on Item 8 of the IRLS (Item 8: When you had RLS symptoms how severe were they on average?)
* At Baseline (Visit 2), subject has a score of ≥ 4 points on the Clinical Global Impression (CGI) Item 1 assessment (indicating moderately ill)

Exclusion Criteria:

* Subject has previously participated in this study or has received previous treatment with Rotigotine
* Subject has participated in another study of an investigational medicinal product (IMP) or a medical device within the last 30 days prior to Visit 1, or is currently participating in another study of an IMP or a medical device
* Subject has secondary RLS (eg, due to Renal Insufficiency [Uremia], Iron Deficiency Anemia or Rheumatoid Arthritis)
* Subject has had a Ferritin value of ≤ 18 µg/L within the last 3 months prior to Baseline (Visit 2)
* Subject has RLS associated with previous or concomitant therapy with Dopamine Receptor Antagonists, Butyrophenones, Metoclopramide, Atypical Antipsychotics (eg, Olanzapine), Tri- and Tetra-Cyclic Antidepressants, Mianserine, or Lithium or H2-Blockers (eg, Cimetidine), or due to withdrawal from drugs such as Anticonvulsants, Benzodiazepines, Barbiturates, and other Hypnotics
* Subject has evidence of an Impulse Control Disorder according to the Modified Minnesota Impulsive Disorders Interview (mMIDI) at Screening (Visit 1)
* Subject has a history of sleep disturbances, such as Sleep Apnea Syndrome (including Obstructive Sleep Apnea), Narcolepsy, Sleep Attacks/Sudden Onset of Sleep, or Myoclonus Epilepsy either observed during Polysomnography (PSG) (local PSG evaluations) or evidenced by subject history
* Subject has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia Suicide Severity Rating Scale (C-SSRS) at Screening (Visit 1)
* Subject has uncontrolled Hypertension according to the judgment of the investigator
* Subject has additional clinically relevant concomitant diseases, such as Attention Deficit Hyperactivity Disorder, Polyneuropathy, Claudication, Varicosis, Muscle Fasciculation, painful legs and moving toes, or Radiculopathy
* Subject has other central nervous system diseases, such as Parkinson's Disease, Dementia, Progressive Supranuclear Paresis, Multisystem Atrophy, Huntington's Chorea, Amyotrophic Lateral Sclerosis, or Alzheimer's Disease
* Subject has a prior history of psychotic episodes
* Subject has a history of chronic alcohol or drug abuse within the last 12 months prior to Visit 1
* Subject has any medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's well being or ability to participate in this study
* Subject has a clinically relevant Venous or Arterial Peripheral Vascular Disease
* Subject has a malignant Neoplastic Disease requiring therapy within 12 months prior to Screening (Visit 1)
* Subject is currently receiving treatment with any of the following drug classes: Neuroleptics, Hypnotics, Antidepressants, Anxiolytic Drugs, Anticonvulsive Therapy, Budipine, Dopamine Antagonist Antiemetics (except Domperidone), Opioids, Benzodiazepines, Monoamine Oxidase (MAO) Inhibitors, Catechol-O-Methyltransferase (COMT) Inhibitors, Sedative Antihistamines, Psychostimulates, or Amphetamines. If subject has received such therapy, a Washout Period of at least 7 days prior to Baseline (Visit 2) is required before starting treatment in this study
* Subject is pregnant, nursing, or is a woman of childbearing potential who is not surgically sterile, 2 years postmenopausal, or does not consistently use 2 combined medically acceptable methods of contraception, including at least 1 barrier method, unless sexually abstinent
* Subject is a shift worker or performs other continuous non-disease-related life conditions which do not allow regular sleep at night
* At Screening Visit (Visit 1) or Baseline Visit (Visit 2), subject has Symptomatic Orthostatic Hypotension with a decrease of Blood Pressure (BP) from supine to standing position of ≥ 20 mmHg in systolic BP or of ≥ 10 mmHg in diastolic BP taken from the 5-minute supine and 1- and/or 3-minute standing measurements at Visit 1 or Visit 2
* Subject is treated with Dopamine Agonists within a period of 7 days prior to Baseline (Visit 2) or L-Dopa within 3 days prior to Baseline (Visit 2)
* Subject has a known history indicating intolerability to prior Dopaminergic therapy (if pretreated) when previously treated with any Dopaminergic agent
* Subject has a known hypersensitivity to any components of the study medication, such as a history of significant skin hypersensitivity to adhesives, known hypersensitivity to other transdermal medications, or has unresolved contact Dermatitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1-877-822-9493
Locations (18):
- United States (18):
  - 006, Birmingham, Alabama
  - 013, Jasper, Alabama
  - 021, Gilbert, Arizona
  - 014, Little Rock, Arkansas
  - 010, Oceanside, California
  - 004, Orange, California
  - 002, Tampa, Florida
  - 012, Macon, Georgia
  - 008, Destrehan, Louisiana
  - 017, Brighton, Massachusetts
  - 016, Brockton, Massachusetts
  - 019, Kalamazoo, Michigan
  - 015, St Louis, Missouri
  - 007, West Seneca, New York
  - 018, Cincinnati, Ohio
  - 009, West Chester, Pennsylvania
  - 003, Austin, Texas
  - 005, San Antonio, Texas

REFERENCES:
- [Derived] Garcia-Borreguero D, Allen R, Hudson J, Dohin E, Grieger F, Moran K, Schollmayer E, Smit R, Winkelman J. Effects of rotigotine on daytime symptoms in patients with primary restless legs syndrome: a randomized, placebo-controlled study. Curr Med Res Opin. 2016;32(1):77-85. doi: 10.1185/03007995.2015.1103216. Epub 2015 Nov 16. PMID 26569149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment for the RL0003 study began in March 2012. It concluded in April 2013. Recruitment for this study took place in the United States of America.
Pre-assignment Details: The participant flow consists of the Randomized Set (RS), which is all subjects randomized into the study.
  The demographics and study outcomes consist of the Full Analysis Set (FAS), which includes all randomized, treated subjects having valid Baseline measurements for both primary efficacy variables.
Groups:
- Rotigotine: Rotigotine patches titrated from 1 mg/ 24 hr - 3 mg / 24 hr or until effective or maximum dose was reached.
  Rotigotine: Transdermal patch containing Rotigotine formulated in an adhesive matrix. Subjects were to be treated with their optimal dose which consisted of one of the dose strengths below:
  Rotigotine 1 mg/ 24 hr, Rotigotine 2 mg/ 24 hr, Rotigotine 3 mg/ 24 hr, One patch every 24 hours
  7 weeks (titration plus maintenance)
Period: Overall Study
Arm/Group | Rotigotine | Placebo
Started | 101 | 49
Completed | 91 | 44
Not Completed | 10 | 5
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Population: The demographics section consists of the Full Analysis Set (FAS), which includes all randomized, treated subjects having valid Baseline measurements for both primary efficacy variables.
Groups:
- Rotigotine: Rotigotine patches titrated from 1 mg/ 24 hr - 3 mg/ 24 hr or until effective or maximum dose was reached.
  Rotigotine: Transdermal patch containing Rotigotine formulated in an adhesive matrix. Subjects were to be treated with their optimal dose which consisted of one of the dose strengths below:
  Rotigotine 1 mg/ 24 hr, Rotigotine 2 mg/ 24 hr, Rotigotine 3 mg/ 24 hr, One patch every 24 hours
  7 weeks (titration plus maintenance)
- Total: Total of all reporting groups
Arm/Group | Rotigotine | Placebo | Total
Number analyzed (Participants) | 101 | 49 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 89 | 44 | 133
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (14.2) | 47.9 (13.7) | 47.9 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 20 | 78
  Male | 43 | 29 | 72
Weight [Mean (Standard Deviation); unit: Kilograms] | 80.93 (15.11) | 80.18 (12.94) | 80.69 (14.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline To The End Of The Maintenance Period in International Restless Legs Scale (IRLS) Sum Score
Description: The International Restless Legs Scale (IRLS) was intended to evaluate, in a standardized way, the subjective intensity of major symptoms of Restless Legs Syndrome (RLS) and, in 2 items (9 and 10), the impact of the disease on subjects functioning in daytime activities by use of a 5-point scale for each of a total of 10 items.
  In all items, the scores ranged from 0 (not present) to 4 (severe). A sum score across all 10 items was calculated for analysis, which varied between 0 (no RLS symptoms present at all) to 40 (maximum severity in all symptoms).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF).
  Out of the 150 patients in the FAS, 150 were included in this analysis.
  The FAS includes all randomized, treated subjects having valid Baseline measurements for both primary efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -15.46 (1.00) | -15.19 (1.29)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; ANCOVA model was used for analysis with fixed effects for treatment assignment (main factor) and the subject's investigational center (stratifying factor) and a covariate for the Baseline Visit value of the IRLS sum score; Test type: Superiority or Other; p = 0.8451, ANCOVA — A hierarchical test procedure was done for the primary efficacy variables at an α-level of 5 %. If a test was statistically significant, a test for the next variable was performed. If a test was not statistically significant the procedure stopped; LS Mean = -0.27, 95% CI 2-sided [-2.96 to 2.42], Standard Error of Mean 1.36

2. Primary Outcome: Change In Average Of Means Of Multiple Suggested Immobilization Test Discomfort Scale (m-SIT-DS) Values Of Each Individual Suggested Immobilization Test (SIT) For The Combination Of Multiple Suggested Immobilization Test (m SIT)
Description: The Multiple Suggested Immobilization Test Discomfort Scale (m-SIT-DS) was used for assessment of the sensory components of Restless Legs Syndrome (RLS) symptoms in order to provide a subjective score of the severity of RLS symptoms during each Suggested Immobilization Test (SIT).
  Scores ranged from 0 (no symptoms) to 10 (very severe symptoms) and were assessed every 10 minutes within each SIT.
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo patches titrated from 1 mg/ 24 hr - 3 mg/ 24 hr or until effective or maximum dose was reached.
  Placebo 1 mg/ 24 hr, Placebo 2 mg/r24 hr, Placebo 3 mg/ 24 hr, one patch every 24 hours
  7 weeks
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -2.83 (0.25) | -2.90 (0.33)
Statistical Analysis 1: Comparison: Rotigotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.8336, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean = 0.07, 95% CI 2-sided [-0.61 to 0.75], Standard Error of Mean 0.34

3. Secondary Outcome: Change In Average Of Means Of Periodic Limb Movement During Wakefulness Index (PLMWI) Change In Average Of Means Of Periodic Limb Movement During Wakefulness Index (PLMWI) For The Combination Of Multiple Suggested Immobilization Test (m-SIT)
Description: During each single Suggested Immobilization Test (SIT) PLMWI was measured using a validated actigraphy device. Simultaneous actigraphy of the legs was performed by an actigraphy device, which was attached to the ankle prior to the start of the SIT. The PLMWI was recorded while the subject was awake.
  Scores ranged from 0 (no symptoms) to 10 (very severe symptoms) and were assessed every 10 minutes within each SIT.
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: Full Analysis Set (FAS) with Last Observation Carried Forward (LOCF).
  Out of the 150 patients in the FAS, 149 were included in this analysis.
  The FAS includes all randomized, treated subjects having valid Baseline measurements for both primary efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 48
units on a scale | -48.05 (6.25) | -56.39 (8.03)

4. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Satisfaction With Sleep (Item 1 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = completely satisfied) to (10 = completely dissatisfied).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -3.44 (0.40) | -3.93 (0.51)

5. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Severity Of Restless Legs Syndrome (RLS) At Bedtime (Item 2 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = none) to (10 = very severe).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -4.62 (0.31) | -4.46 (0.40)

6. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Severity Of Restless Legs Syndrome (RLS) During The Night (Item 3 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = none) to (10 = very severe).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -4.46 (0.29) | -4.45 (0.38)

7. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Severity Of Restless Legs Syndrome (RLS) At Daytime At Rest (Item 4 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = none) to (10 = very severe).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -3.44 (0.27) | -2.94 (0.35)

8. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Severity of Restless Legs Syndrome (RLS) At Daytime In Activity (Item 5 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = none) to (10 = very severe).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -1.80 (0.21) | -1.69 (0.27)

9. Secondary Outcome: Change In Item Score From Baseline To The End Of The Maintenance Period In Daytime Tiredness (Item 6 of Restless Legs Syndrome 6 Rating Scales [RLS-6])
Description: The RLS-6 is an 11-point scale. This 11-point scale was provided with ranges between (0 = not at all) to (10 = very severe).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -3.02 (0.31) | -3.09 (0.40)

10. Secondary Outcome: Change From Baseline To The End Of Maintenance Period In Daytime Somnolence Domain Score Of The Medical Outcomes Study (MOS) Sleep Scale - Revised (MOS Sleep-R)
Description: The Medical Outcomes Study (MOS) Sleep Scale-Revised (MOS Sleep-R) is a self-administered questionnaire measuring several important aspects of sleep that have been validated in both general and patient populations.
  The MOS Sleep-R consists of 12-items. Responses for 10 of the 12 items are on a 5-point frequency scale with options ranging from "all of the time" to "none of the time". The other two items ask about the length of time to fall asleep and the average number of hours slept per night. The sleep problems index I allows for the summary of sleep problems using an abbreviated six-item index, whereas the sleep problems index II uses nine of the 12 items of the scale to compute an overall sleep problem summary. A higher score on each scale in summary index represents a lack of sleep problems (better sleep quality). All scores are transformed linearly to range from 0 to 100, with the exception of the sleep quantity subscale, which is scored in hours.
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 15.28 (2.30) | 14.05 (2.95)

11. Secondary Outcome: Change From Baseline To The End of Maintenance Period In Sleep Disturbance Domain Score Of The Medical Outcomes Study (MOS) Sleep Scale - Revised (MOS Sleep-R)
Description: as for outcome 10
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 30.29 (2.82) | 29.10 (3.60)

12. Secondary Outcome: Change From Baseline To The End of Maintenance Period In Sleep Adequacy Domain Score Of The Medical Outcomes Study (MOS) Sleep Scale - Revised (MOS Sleep-R)
Description: as for outcome 10
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo patches titrated from 1 mg/ 24 hr - 3 mg/r24 hr or until effective or maximum dose was reached.
  Placebo 1 mg/ 24 hr, Placebo 2 mg/ 24 hr, Placebo 3 mg/ 24 hr, one patch every 24 hours
  7 weeks
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 23.40 (3.09) | 22.88 (3.96)

13. Secondary Outcome: Change From Baseline To The End of Maintenance Period In Sleep Quantity Domain Score Of The Medical Outcomes Study (MOS) Sleep Scale - Revised (Sleep Scale-R)
Description: as for outcome 10
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 0.87 (0.17) | 1.11 (0.21)

14. Secondary Outcome: Change In Total Score From Baseline To The End of Maintenance Period On Profile Of Mood States Questionnaire (POMS)
Description: The Profile of Mood States questionnaire (POMS) total score will be calculated as the sum of the scores for the following 5 scale scores (Tension-Anxiety, Depression-Dejection, Anger-Hostility, Fatigue-Inertia, and Confusion-Bewilderment) and then subtracting the Vigor-Activity score. All factors have to be available for the total score to be calculated; otherwise the total score will be set to missing. The range for the POMS is 0 - 200 with a high score being negative and a low score being positive.
  For the POMS questionnaire total score, descriptive statistics will be presented on both the observed and the change from Baseline to the end of the Maintenance Period values for the Full Analysis Set (FAS).
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | -8.27 (3.01) | -9.07 (3.80)

15. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary Score
Description: The SF-36 is a 36 item generic human research quality of life instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and a further unscaled single item (question 2) for perceived stability or change in health (Health Transition) during the last year. The norm-based scores (based on the US general population) were used for analysis. For the MCS, the lowest and highest possible scores are -9 and 82 (rounded).
  The SF-36 domains (subscores) are scored so that a higher score indicates a better health state.
Time Frame: Baseline to End of Maintenance Period (approximately 7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 1.77 (1.01) | 1.79 (1.29)

16. Secondary Outcome: Change From Baseline in SF-36 Physical Component Summary Score
Description: The SF-36 is a 36 item generic human research quality of life instrument that uses a recall period of 4 weeks. Items are grouped into 8 domains as follows: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items), and a further unscaled single item (question 2) for perceived stability or change in health (Health Transition) during the last year. The norm-based scores (based on the US general population) were used for analysis. For the PCS, the lowest and highest possible scores are 1 and 81 (rounded).
  The SF-36 domains (subscores) are scored so that a higher score indicates a better health state.
Time Frame: Baseline to End of Maintenance Period (7 weeks)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Rotigotine | Placebo
Number analyzed (Participants) | 101 | 49
units on a scale | 2.16 (0.76) | 2.28 (0.98)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded during the course of the RL0003 study, which began in March 2012 and concluded in April 2013.
Description: Adverse Event reporting consists of the Safety Set (SS). The SS consists of all randomized subjects that received at least 1 dose of study drug.
Arm/Group | Rotigotine | Placebo
Serious Adverse Events (participants affected / at risk) | 2/101 | 0/49
Other Adverse Events (participants affected / at risk) | 42/101 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=101) | Placebo (N=49)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotigotine (N=101) | Placebo (N=49)
Nausea (Gastrointestinal disorders) | 16 (19) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Application site pruritus (General disorders) | 12 (15) | 2 (2)
Headache (Nervous system disorders) | 10 (13) | 5 (9)
Somnolence (Nervous system disorders) | 8 (9) | 4 (4)
Dizziness (Nervous system disorders) | 8 (8) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.